CLINICAL TRIAL: NCT04512443
Title: Clinical Efficacy of Conservative Treatment in Female Patients With Plevic Congestion Syndrome
Status: Completed | Type: Observational
Sponsor: Interregional Clinical Diagnostic Center, Russia (Other)
Responsible Party: Principal Investigator, Akhmetzianov Rustem, Principal Investigator, Interregional Clinical Diagnostic Center, Russia
Other Study IDs: Daflon25122019
Record Dates: First submitted 2020-08-10; First posted 2020-08-13 (Actual); Last update posted 2020-08-13 (Actual); Status verified 2020-08

CONDITIONS: Pelvic Congestion Syndrome
MeSH Terms: interventions — Diosmin

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 1: 42 women (treated with Daflon 1000 mg (study group))
  Interventions: Drug: Daflon
- 2: 41 women (placebo (control group))

INTERVENTIONS:
Drug: Daflon — All consecutive patients were randomly allocated into 2 groups to receive Daflon (Detralex) at a dose of 1000 mg once daily (study group) or placebo (control group).
  Groups: 1

SUMMARY:
The article presents the results of a randomized, placebo-controlled study of the conservative treatment with Daflon (Detralex) in female patients with Pelvic congestion syndrome .

ELIGIBILITY:
Inclusion Criteria:

•The presence of pelvic varicose veins verified by transvaginal and transabdominal duplex ultrasound scanning

Exclusion Criteria:

* Severe disease of the gastrointestinal tract or hematopoietic system
* Terminal stage of cardiovascular, respiratory, renal or hepatic failure
* Grade IV malignancy
* Peripheral artery disease (PAD) of the lower extremities, any type of diabetes, or mental disease.
* Pregnant women at any gestational age, women who gave birth less than 12 months ago, and breastfeeding mothers.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: women with Pelvic congestion syndrome
Sampling Method: Non-Probability Sample
Enrollment: 83 (Actual)
Dates: Start 2019-12-28 (Actual); Primary Completion 2020-03-28 (Actual); Study Completion 2020-03-28 (Actual)

PRIMARY OUTCOMES:
Pelvic Varicose Veins Questionnaire | 2 months
  Assessment of quality of life according to the questionnaire before and after treatment

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Akhmetzianov Rustem, Kazan'
  - Roman Bredikhin, Kazan'